CLINICAL TRIAL: NCT04208308
Title: Comparison of Effect of Animal and Plant Sources of Omega-3 PUFA in Prevention of Cardiovascular and Metabolic Diseases
Brief Title: Omega-3 PUFA in Prevention of Cardiovascular and Metabolic Diseases (CARDMET3)
Acronym: CARDMET3
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pavol Jozef Safarik University (Other)
Responsible Party: Principal Investigator, Martin Janičko, Assistant professor, Pavol Jozef Safarik University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UEM001LFPJSU
Record Dates: First submitted 2019-11-06; First posted 2019-12-23 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Obesity, Abdominal; Metabolic Syndrome; Cardiovascular Risk Factor
MeSH Terms: conditions — Obesity, Abdominal; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Healthy and obese people in different age categories.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Control negative group (No Intervention): Without supplementation
- Experimental negative group I (Experimental): Chia seeds supplementation (25 g)
  On dose (25g) of chia seeds contains:
  energy 498,75 kJ / 118,75 kcal, protein 3,25 g, carbohydrates 9 g, fiber 6 g, fats 6,5 g, Calcium 160 mg Phosphorus 247,5 mg Kalium 37,5 mg Natrium 5,25 mg Zincum 0,975 mg Manganum 0,625 mg Omega-3 fatty acids 4,475 g Omega-6 fatty acids 1,475 g Vitamin B1 0,1 mg Vitamin B2 0,0075 mg Vitamin B3 0,75 mg Vitamin C 0,2 mg
  Interventions: Dietary Supplement: Chia seeds supplementation (25 g)
- Experimental negative group II (Experimental): Chia seeds supplementation (15 g)
  On dose (15g) of chia seeds contains:
  energy 299 kJ / 71,2 kcal, protein 1,95 g, carbohydrates 5,4 g, fiber 3,6 g, fats 3,9 g, Calcium 96 mg Phosphorus 148,5 mg Kalium 22,5 mg Natrium 3,15 mg Zincum 0,59 mg Manganum 0,375 mg Omega-3 fatty acids 2,684 g Omega-6 fatty acids 0,885 g Vitamin B1 0,06 mg Vitamin B2 0,0045 mg Vitamin B3 0,45 mg Vitamin C 0,12 mg
  Interventions: Dietary Supplement: Chia seeds supplementation (15 g)
- Experimental negative group III (Experimental): Combine supplementation: chia seeds and fish oil
  Daily dose:
  Chia seeds supplementation (15 g) and fish oil supplementation (pharmacological supplement) - Maxi Cor 70+20 (EPA 675 mg +DHA 510 mg)
  On dose (15g) of chia seeds contains:
  energy 299 kJ / 71,2 kcal, protein 1,95 g, carbohydrates 5,4 g, fiber 3,6 g, fats 3,9 g, Calcium 96 mg Phosphorus 148,5 mg Kalium 22,5 mg Natrium 3,15 mg Zincum 0,59 mg Manganum 0,375 mg Omega-3 fatty acids 2,684 g Omega-6 fatty acids 0,885 g Vitamin B1 0,06 mg Vitamin B2 0,0045 mg Vitamin B3 0,45 mg Vitamin C 0,12 mg
  Interventions: Dietary Supplement: Combine supplementation: chia seeds (15g) and fish oil Maxi Cor 70+20
- Experimental negative group IV (Experimental): Fish oil supplementation
  Daily dose:
  Fish oil supplementation (pharmacological supplemment) - Maxi Cor 70+20 (EPA 825 mg +DHA 525 mg)
  Interventions: Dietary Supplement: Fish oil supplementation
- Control positive group (No Intervention): Without supplementation
- Experimental positive group I (Experimental): Chia seeds supplementation (25 g)
  On dose (25g) of chia seeds contains:
  energy 498,75 kJ / 118,75 kcal, protein 3,25 g, carbohydrates 9 g, fiber 6 g, fats 6,5 g, Calcium 160 mg Phosphorus 247,5 mg Kalium 37,5 mg Natrium 5,25 mg Zincum 0,975 mg Manganum 0,625 mg Omega-3 fatty acids 4,475 g Omega-6 fatty acids 1,475 g Vitamin B1 0,1 mg Vitamin B2 0,0075 mg Vitamin B3 0,75 mg Vitamin C 0,2 mg
  Interventions: Dietary Supplement: Chia seeds supplementation (25 g)
- Experimental positive group II (Experimental): Chia seeds supplementation (15 g)
  On dose (15g) of chia seeds contains:
  energy 299 kJ / 71,2 kcal, protein 1,95 g, carbohydrates 5,4 g, fiber 3,6 g, fats 3,9 g, Calcium 96 mg Phosphorus 148,5 mg Kalium 22,5 mg Natrium 3,15 mg Zincum 0,59 mg Manganum 0,375 mg Omega-3 fatty acids 2,684 g Omega-6 fatty acids 0,885 g Vitamin B1 0,06 mg Vitamin B2 0,0045 mg Vitamin B3 0,45 mg Vitamin C 0,12 mg
  Interventions: Dietary Supplement: Chia seeds supplementation (15 g)
- Experimental positive group III (Experimental): Combine supplementation: chia seeds and fish oil
  Daily dose:
  Chia seeds supplementation (15 g) and fish oil supplementation (pharmacological supplement) - Maxi Cor 70+20 (EPA 675 mg +DHA 510 mg)
  On dose (15g) of chia seeds contains:
  energy 299 kJ / 71,2 kcal, protein 1,95 g, carbohydrates 5,4 g, fiber 3,6 g, fats 3,9 g, Calcium 96 mg Phosphorus 148,5 mg Kalium 22,5 mg Natrium 3,15 mg Zincum 0,59 mg Manganum 0,375 mg Omega-3 fatty acids 2,684 g Omega-6 fatty acids 0,885 g Vitamin B1 0,06 mg Vitamin B2 0,0045 mg Vitamin B3 0,45 mg Vitamin C 0,12 mg
  Interventions: Dietary Supplement: Combine supplementation: chia seeds (15g) and fish oil Maxi Cor 70+20
- Experimental positive group IV (Experimental): Fish oil supplementation
  Daily dose:
  Fish oil supplementation (pharmacological supplemment) - Maxi Cor 70+20 (EPA 825 mg +DHA 525 mg)
  Interventions: Dietary Supplement: Fish oil supplementation

INTERVENTIONS:
Dietary Supplement: Chia seeds supplementation (25 g) — Dosage: 1 daily dose energy 498,75 kJ / 118,75 kcal, protein 3,25 g, carbohydrates 9 g, fiber 6 g, fats 6,5 g, Calcium 160 mg Phosphorus 247,5 mg Kalium 37,5 mg Natrium 5,25 mg Zincum 0,975 mg Manganum 0,625 mg Omega-3 fatty acids 4,475 g Omega-6 fatty acids 1,475 g Vitamin B1 0,1 mg Vitamin B2 0,0075 mg Vitamin B3 0,75 mg Vitamin C 0,2 mg
  Arms: Experimental negative group I; Experimental positive group I
Dietary Supplement: Chia seeds supplementation (15 g) — Dosage: 1 daily dose energy 299 kJ / 71,2 kcal, protein 1,95 g, carbohydrates 5,4 g, fiber 3,6 g, fats 3,9 g, Calcium 96 mg Phosphorus 148,5 mg Kalium 22,5 mg Natrium 3,15 mg Zincum 0,59 mg Manganum 0,375 mg Omega-3 fatty acids 2,684 g Omega-6 fatty acids 0,885 g Vitamin B1 0,06 mg Vitamin B2 0,0045 mg Vitamin B3 0,45 mg Vitamin C 0,12 mg
  Arms: Experimental negative group II; Experimental positive group II
Dietary Supplement: Combine supplementation: chia seeds (15g) and fish oil Maxi Cor 70+20 — Chia seeds - 1 daily dose Fish oil TID
  Chia seeds supplementation (15 g) and fish oil supplementation (pharmacological supplement) - Maxi Cor 70+20 (EPA 675 mg +DHA 510 mg)
  On dose (15g) of chia seeds contains:
  energy 299 kJ / 71,2 kcal, protein 1,95 g, carbohydrates 5,4 g, fiber 3,6 g, fats 3,9 g, Calcium 96 mg Phosphorus 148,5 mg Kalium 22,5 mg Natrium 3,15 mg Zincum 0,59 mg Manganum 0,375 mg Omega-3 fatty acids 2,684 g Omega-6 fatty acids 0,885 g Vitamin B1 0,06 mg Vitamin B2 0,0045 mg Vitamin B3 0,45 mg Vitamin C 0,12 mg
  Arms: Experimental negative group III; Experimental positive group III
Dietary Supplement: Fish oil supplementation — TID
  Daily dose:
  Fish oil supplementation (pharmacological supplemment) - Maxi Cor 70+20 (EPA 825 mg +DHA 525 mg)
  Arms: Experimental negative group IV; Experimental positive group IV

SUMMARY:
The study is aimed to assess the efficacy of animal, plant sources of omega-3 polyunsaturated fatty acids and omega-3 pharmacological supplements on obesity, metabolic syndrome and cardiovascular disease.

DETAILED DESCRIPTION:
More than four million people in Europe (47%) and more than 1.9 million people in European Union (EU) (40%) die of cardiovascular diseases (CVD) every year. CVD mortality in EU is 43% in women and 36% in men. In Central and Eastern Europe, much more people die of CVD than in Western, Northern and Southern European countries. The World Health Organization (WHO) states that number of deaths in Slovakia is much higher than in Western European countries, even higher than in V4 countries - Slovakia, Czech Republic, Poland and Hungary

In the first stage of the project fatty acids will be analyzed with the focus on the ratio of omega-6 and omega-3 polyunsaturated fatty acids in fatty food for normal consumption and in nutritional supplements containing omega-3 polyunsaturated fatty acids.

In the second phase of the project risk factors of cardiovascular diseases for people without and people with a history of cardiovascular disease will be monitored and compared. There will be monitored and compared a wide range of laboratory markers of clinical biochemistry, immunology, pathological physiology in order to determine cardiovascular risk for men and women in different age categories.

The third stage will monitor the effect of natural plant and animal sources and pharmacological nutritional supplements with omega-3 polyunsaturated fatty acids on obesity, metabolic syndrome and cardiovascular risk factors.

The aim of this study is to assess the efficacy of animal, plant sources of omega-3 polyunsaturated fatty acids and omega-3 pharmacological supplements on obesity, metabolic syndrome and cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* for obese participants were BMI≥29, age ≥18 and non-smokers, cardiovascular diseases. metabolic syndrome, obesity
* for healthy participants with normal weight, inclusion criteria BMI25, age ≥18, non-smokers

Exclusion Criteria:

* for all participants were cancer, inflammatory diseases, tuberculosis, renal and hepatic insufficiency, and pregnancy
* for healthy participants without cardiovascular diseases, obesity and metabolic syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-01-15 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Body mass index | 6 months
  BMI kg/m2 6 months change.
glucose levels | 6 months
  fasting glucose in mmoL/L
Change in total cholesterol from baseline | 6 months
  percentual change in total cholesterol (mmoL/L) from baseline to 6months followup
  - total genetic analysis, extracellular DNA
Systemic inflammation activity | 1 months
  Interleukin 1 levels, interleukin 6 levels (pg/mL)
Antioxidant status | 18 months
  Determination of total antioxidant capacity (mmoL/L)
Change in estrogen concentration | 6 months
  Assesment of concentration of estrogen (ng/mL)
Bile acids in serum | 6 months
  Concentration of serum bile acids (pg/mL)
Tissue concentrations of nitric oxide | 6months
  Determination of nitric oxide synthetase activity by electron microscopy
NF kappa B activity | 6 months
  Determination of NF kappa B activity by electron microscopy
Catalase activity | 6 months
  Determination of Catalase activity by electron microscopy
Superoxide dismutase activity | 6 months
  Determination of Superoxide dismutase activity by electron microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Zdenka Hertelyová, Dr., PhD., Study Director — Pavol Josef Šafarik University, Faculty of Medicine, 040 11 Košice, Slovakia
Locations (1):
- 1st Department of Internal medicine, L. Pasteur University Hospital in Košice, Košice, Slovakia

IPD SHARING:
Plan to Share IPD: No